CLINICAL TRIAL: NCT05993910
Title: Prospektive Hyperthermie-Datenbank Bei Krebspatienten (HTRegister)
Brief Title: Prospective Hyperthermia Database in Cancer Patients (HT Register)
Acronym: HTRegister
Status: Recruiting | Type: Observational
Sponsor: Pirus Ghadjar (Other)
Responsible Party: Sponsor-Investigator, Pirus Ghadjar, Prof. Dr. med., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: HTRegister2014
Record Dates: First submitted 2023-08-03; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Hyperthermia; Cancer
Keywords: Hyperthermia E02.565; HTRegister
MeSH Terms: conditions — Hyperthermia; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Blood and tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hyperthermie Register: Hyperthermia simultaneous with Radiotherapy alone, Hyperthermia simultaneous with Chemotherapy alone, Hyperthermia simultaneous with Radiochemotherapy alone
  Interventions: Other: Hyperthermie Register

INTERVENTIONS:
Other: Hyperthermie Register — * die Höhe der Temperatur im Zielgebiet (42,5 bis 43 °C),
  * die Dauer der Anwendung und
  * die simultane Therapie mit Chemo- und/oder Strahlentherapie

SUMMARY:
This monocentric study registry records all cancer patients at the Charité which are treated with hyperthermia to examine the therapeutic use of hyperthermia in cancer patients in the general application and to obtain an accurate risk-benefit balance

After confinement in this database are the patients prospectively in order to complications, disease status and survival status tracked.

Furthermore there is the possibility in the course of this study to an optional take part in translational accompanying research with the aim of prognostic factors for response to hyperthermia treatment.

DETAILED DESCRIPTION:
A total of 1000 patients with various diseases with the indication for hyperthermia in addition to standard oncological therapy (radiation therapy, chemotherapy, radiochemotherapy) will be included in this registry protocol.

ELIGIBILITY:
Inclusion Criteria:

* Contrazeption with female patients at the capable of bearing children age
* Written agreement is present (DvH, ICH-GCP)
* Patients, who participate at the same time in a interventional study, can nevertheless in this register study participate if this none Exclusion criterion for the interventional study represents.
* With children must the treatment with one of the GPOH agreed Pattern take place

Exclusion Criteria:

* Exclusion criteria for the hyperthermia (such as hip prosthesis in the therapeutic area, metal implants/marker, patients with cardiac pacemakers)
* mental disease, what the proper study participation does not allow.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It is planned to include the first 1.000 patients in this prospective database. Because of the characters in the database is a certain gender distribution not laid down . Confinement are capable of all patients in the Charité , which has a hyperthermia treatment , regardless of age or gender
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Effectivity | Through the study completion, up to 10 years
  To determine the effectiveness of hyperthermia treatment, patients are tracked in terms of overall survival , progression-free survival and disease-free survival
Toxicity | Through the study completion, up to 10 years
  Toxicity assessment based on Common Toxicity Criteria Scoring

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Radio - Oncology and Radiotherapy, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes